CLINICAL TRIAL: NCT01255436
Title: Effectiveness of SMS Text Reminders to Improve Blood Pressure Among Patients With Hypertension at a General Medicine Outpatient Clinic in a Tertiary Center in Manila, Philippines: A Randomized Controlled Trial
Brief Title: Effectiveness of SMS Text Reminders to Improve Blood Pressure Among Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Philippines (Other)
Collaborators: Department of Health, Philippines (Other Government)
Responsible Party: Principal Investigator, Lia M. Palileo, Clinical Associate Professor, University of the Philippines
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCS IM 2010-002 (R-006TE)
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS text reminders (Experimental): Participants in this arm will receive SMS text messages on top of the usual care they receive from their physicians.
  Interventions: Other: SMS text reminders
- Usual Care (Other): Participants in this arm will receive the usual care they receive from their physicians.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: SMS text reminders — Patients in the intervention arm will receive 2 text messages per week delivered via SMS on randomly chosen days and times during the 12-week study period. The aims of the messages are to remind patients to take their blood pressure medications daily, what the target blood pressure is, and the benefits of daily intake of anti-hypertensive medications.
  Arms: SMS text reminders
Other: Usual Care — Patients in the usual care arm will receive the care usually provided by their physicians. This consists of consultations, medical advice, and prescriptions for maintenance medications. They will not be sent any SMS text reminders from the study.
  Other Names: No SMS text reminders
  Arms: Usual Care

SUMMARY:
Objective: To test the primary hypothesis that SMS text messages delivered to patients via mobile phone can improve blood pressure within 12 weeks compared to usual care

Design: Parallel group, randomized, controlled trial; the patient is the unit of randomization

Setting: General Medicine Outpatient Continuity Clinic of the Philippine General Hospital and Private Outpatient Clinics near the Philippine General Hospital

Patients: Ambulatory men and women aged 19 years and older (N=700) with a diagnosis of essential hypertension, on maintenance blood pressure-lowering medications, who have daily access to a mobile phone in the household and know or live with someone who knows how to retrieve, read and reply to text messages using a mobile phone

Intervention: SMS text messages delivered twice a week for 12 weeks, which aim to 1) provide information regarding hypertension; 2) remind patients to take their medications.

Main Outcome Measure: The primary outcomes are the mean change in systolic and diastolic blood pressures at the end of 12 weeks. The secondary outcomes are improvement in blood pressure control rate and medication adherence.

DETAILED DESCRIPTION:
The study will be done in 2 phases:

Phase I: Development of the SMS text messages

The SMS messages to be used in the trial will be developed and pre-tested in focus group discussions of a convenience sample of subjects similar to the target population for understandability and acceptability.

Phase II: Parallel group, open-label, randomized, controlled trial

Target Population

Hypertensive patients being seen at the General Medicine Outpatient Clinic of a public, tertiary, university hospital in Manila, Philippines

Sampling Method

A criterion sampling strategy will be used in the study. Patients who fulfill the eligibility criteria will be recruited consecutively until the desired sample size is reached.

Randomization and Allocation Concealment

Eligible patients will be randomized to one of two treatment groups using a computer-generated random allocation sequence. Allocation of treatment will be done by a third party using sequential, sealed opaque envelopes.

Blinding

Given the nature of the intervention, patients will not be blinded to the treatment groups. However, measures will be taken to blind the physicians managing the participants at the clinic. Outcome assessors will also be blinded to the participants' treatment groups.

Procedures and Measurements

Written, informed consent will be obtained prior to enrolment in the study. Once an eligible participant has given consent, he will be randomized to either the intervention or control arm of the trial by a third party using sequentially numbered opaque envelopes. At the end of a 12-week follow up period, participants will be asked to return for a final study visit, where blood pressure and medication adherence will be measured. Acceptability of the SMS intervention will also be determined using a structured questionnaire. A period of four weeks from scheduled date of final visit is allowed before a patient is considered to have been lost to follow-up.

Intervention: SMS reminders

Patients in the intervention arm will receive 2 text messages per week delivered via SMS on randomly chosen days and times during the 12-week study period. The aims of the messages are to remind patients to take their blood pressure medications daily, what the target blood pressure is, and the benefits of daily intake of anti-hypertensive medications. Successful contact will be assumed when "Message sent" is seen on the screen. Otherwise, the same text message shall be immediately resent up to a maximum of 3 times. Receipt of the messages will be free to the study participants and independent of their telephone service provider.

Control: Usual Care

Routine or usual care of hypertensive patients at the General Medicine Outpatient clinic is based on the Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. This consists of physician visits, advice and medication prescription by the healthcare provider. It does not include sending SMS messages to encourage adherence and provide information regarding hypertension.

Outcome Measurements

Blood Pressure

Blood pressure will be measured using a calibrated digital sphygmomanometer manufactured by Omron after the participant has been seated quietly for five minutes. The average of two readings taken five minutes apart will be recorded.

Medication Adherence

The Adherence Self-Report Questionnaire (ASRQ), a brief, validated, self-administered questionnaire, will be used to measure medication adherence. Participants will be asked to complete the Filipino translation of the ASRQ.

Acceptability of SMS Messages

Acceptability of the SMS messages will be measured using a brief, self-administered questionnaire.

Planned Analysis

Descriptive statistics for baseline characteristics, adherence scores, and adherence rates in both groups (mean, sd, frequency (%), median) will be computed. Between-group comparisons will be done at baseline to check for similarity of baseline characteristics, and at the end of 12 weeks to test the hypothesis of inequality between two populations. All hypothesis tests will be one-sided with a level of significance set at 0.05. Intention-to-treat (ITT) analysis will be done, with possible sensitivity analysis for drop-outs. All statistical computations will be computed using the Stata statistical software.

Sample Size

The NCSS-PASS statistical software was used to compute for the desired sample size.

The sample size required to fulfill the objectives of the study is 286 subjects per group. Allowing for a loss to follow up of approximately 20%, the final sample size is 350 subjects per group (total of 700 subjects).

Ethical Considerations

Ethics approval will be obtained prior to conducting this study. Written informed consent will be obtained from all participants prior to enrolment. Good clinical practice guidelines will be followed during the course of the study.

At the beginning of the trial, it will be emphasised that communication through SMS in this study is one-way (provider to patient), so there will be no reply to any and all text messages received from participants. The participants will also be advised to consult their physicians for any problems they may experience.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult patients of both sexes with age at least 19 years old being seen at the General Medicine Outpatient Clinic of the Philippine General Hospital
* A diagnosis of hypertension in the medical record
* On at least 1 maintenance medication for hypertension for at least 1 month
* A systolic blood pressure greater than 129 mmHg and less than 160 mmHg or a diastolic blood pressure greater than 79 mmHg or less than 100 mmHg at the time of screening
* Patients with daily access to a mobile phone in the household
* Patients who live with someone who knows how to retrieve and read text messages on their mobile phone, and can relay these messages to them
* Written informed consent

Exclusion Criteria:

* Participation in other studies within one month of trial initiation
* Patients who are unable or refuse to give informed consent
* Patients who have a clinical condition that might interfere with the study (dementia, psychological disorder)
* Patients who share a household with another patient who has already been recruited to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lia M. Palileo, MD, Principal Investigator — University of the Philippines Manila
Locations (1):
- Philippine General Hospital, Manila, Philippines

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with hypertension, maintained on blood pressure-lowering medications, who fulfilled the inclusion/exclusion criteria, and consulting at the General Medicine outpatient continuity clinic were recruited over a period of 6 months.
Groups:
- SMS Text Reminders: 2 SMS text reminders per week for 12 weeks
- No SMS Text Reminders: Usual care consisting of clinic visits, physician advice and medication prescriptions
Period: Overall Study
Arm/Group | SMS Text Reminders | No SMS Text Reminders
Started | 333 (350 patients enrolled but 17 excluded because of missing baseline data.) | 329 (350 patients enrolled but 21 excluded because of missing baseline data)
Completed | 151 | 135
Not Completed | 182 | 194
Not completed — Lost to Follow-up | 178 | 191
Not completed — Death, stroke, or MI | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMS Text Reminders | No SMS Text Reminders | Total
Number analyzed (Participants) | 333 | 329 | 662
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.7) | 59.6 (11.1) | 59.3 (10.9)
Gender [Count of Participants; unit: Participants]
  Female | 220 | 212 | 432
  Male | 113 | 117 | 230
Employment Status [Number; unit: participants]
  Unemployed | 242 | 238 | 480
  Employed | 70 | 65 | 135
  Retired | 21 | 26 | 47
Educational Attainment [Number; unit: participants]
  No formal education | 0 | 2 | 2
  Elementary | 84 | 79 | 163
  High school | 145 | 152 | 297
  College | 89 | 82 | 171
  Other | 15 | 14 | 29
Time in years since diagnosis of hypertension [Mean (Standard Deviation); unit: years] | 8.5 (11.1) | 8.6 (8.2) | 8.5 (10.4)
Number of prescribed drugs for hypertension [Median (Full Range); unit: medications] | 2 [1 to 5] | 2 [1 to 4] | 2 [1 to 5]
Number of prescribed maintenance medications [Median (Full Range); unit: medications] | 3 [1 to 10] | 4 [1 to 13] | 4 [1 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Change in Systolic Blood Pressure After 12 Weeks
Description: Absolute change in systolic blood pressure from baseline to 12 weeks
Time Frame: baseline and 12 weeks
Population: Only participants who completed follow up and had evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SMS Text Reminders | No SMS Text Reminders
Number analyzed (Participants) | 151 | 135
mmHg | -13.7 (19.1) | -9.5 (25.7)
Statistical Analysis 1: Comparison: SMS Text Reminders vs No SMS Text Reminders; Test type: Superiority or Other; p = 0.06, t-test, 1 sided — p-value<0.05 is considered significant; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-9.4 to 1.0]

2. Primary Outcome: Mean Absolute Change in Diastolic Blood Pressure After 12 Weeks
Description: Absolute change in diastolic blood pressure from baseline to 12 weeks
Time Frame: baseline and 12 weeks
Population: Only patients who completed follow up and had evaluable data were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SMS Text Reminders | No SMS Text Reminders
Number analyzed (Participants) | 151 | 135
mmHg | -6.2 (11.1) | -4.7 (12.3)
Statistical Analysis 1: Comparison: SMS Text Reminders vs No SMS Text Reminders; Test type: Superiority or Other; p = 0.14, t-test, 1 sided — p-value < 0.05 considered significant; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.1 to 1.3]

3. Secondary Outcome: Medication Adherence Rate
Description: The percentage of patients with an improvement of at least one point in adherence score as measured by the Adherence Self-Report Questionnaire at the end of 12 weeks Scale Range: 1 to 6, with 1 being the highest (most adherent) and 6 being the lowest (least adherent)
Time Frame: 12 weeks
Population: Only patients who completed follow up and had evaluable data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SMS Text Reminders | No SMS Text Reminders
Number analyzed (Participants) | 151 | 135
percentage of participants | 59.6 | 47.4
Statistical Analysis 1: Comparison: SMS Text Reminders vs No SMS Text Reminders; Test type: Superiority or Other; p = 0.045, Fisher Exact; Risk Ratio (RR) = 1.3, 95% CI 2-sided [1.0 to 1.6] — Numerator is Treatment Group (SMS reminders) and Denominator is Control Group (No SMS reminders)

4. Secondary Outcome: Percentage of Patients With Controlled Blood Pressure at the End of 12 Weeks
Description: The percentage of patients with systolic blood pressure less than 140 mmHg and diastolic blood pressure less than 90 mmHg at the end of 12 weeks
Time Frame: 12 weeks
Population: Only patients who completed follow up and had evaluable data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SMS Text Reminders | No SMS Text Reminders
Number analyzed (Participants) | 151 | 135
percentage of participants | 68.2 | 54.1
Statistical Analysis 1: Comparison: SMS Text Reminders vs No SMS Text Reminders; Test type: Superiority or Other; p = 0.014, Fisher Exact; Risk Ratio (RR) = 1.3, 95% CI 2-sided [1.04 to 1.53]

ADVERSE EVENTS:
Arm/Group | SMS Text Reminders | No SMS Text Reminders
Serious Adverse Events (participants affected / at risk) | 4/333 | 3/329
Other Adverse Events (participants affected / at risk) | 0/333 | 0/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SMS Text Reminders (N=333) | No SMS Text Reminders (N=329)
All-cause mortality (General disorders) | 3 (3) | 2 (2) — Cause of death unspecified.
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Strong conclusions cannot be made because of the high attrition rate at the end of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes